CLINICAL TRIAL: NCT02448628
Title: A Multi-center, Open Label, Dose Titration, Exploratory Study to Evaluate Efficacy and Safety of CS-3150 in Japanese Hypertensive Patients With Moderate Renal Impairment.
Brief Title: A Phase 2 Exploratory Study of CS-3150 in Japanese Hypertensive Patients With Moderate Renal Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS3150-A-J206
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Hypertension
Keywords: Hypertension; moderate renal impairment; mineralocorticoid receptor antagonist; CS-3150; Japanese
MeSH Terms: conditions — Hypertension | interventions — esaxerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CS-3150 (Experimental): CS-3150 1.25 to 5.0 mg , orally, once daily after breakfast for 12 weeks
  Interventions: Drug: CS-3150

INTERVENTIONS:
Drug: CS-3150

SUMMARY:
This study is a multi-center, open label, dose titration, exploratory study to evaluate efficacy and safety of CS-3150 in Japanese hypertensive patients with moderate renal impairment. Primary endpoint is change from baseline in sitting systolic and diastolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Men and women Aged 20 years or older and 80 years or younger at informed consent
* Subjects with hypertension (Sitting systolic blood pressure SBP >= 140 mmHg and < 180 mmHg, Sitting diastolic blood pressure DBP >= 80 mmHg and < 110 mmHg)
* estimated glomerular filtration rate eGFR >= 30 mL/min/1.73 m2 and < 60 mL/min/1.73 m2

Exclusion Criteria:

* Secondary hypertension or malignant hypertension
* Diabetes mellitus with albuminuria
* Serum potassium level < 3.5 or >= 5.1 mEq/L
* Subjects under Insulin treatment
* Subjects under or pre-planned for hemodialysis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sitting systolic and diastolic blood pressure | Baseline to end of Week 12

SECONDARY OUTCOMES:
Change from baseline in UACR | Baseline to end of Week 12
  Urine Albumin Creatinine Ratio (UACR)

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/